CLINICAL TRIAL: NCT02870608
Title: Interest of Measuring Lung Elasticity ELASTOgraphy in the Fetus in the Case of PreMAture Childbirth Threat
Acronym: ELASTOMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: API/2015/60
Record Dates: First submitted 2016-07-21; First posted 2016-08-17 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy Complications; Obstetric Labor, Premature
Keywords: Elastography
MeSH Terms: conditions — Pregnancy Complications; Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preterm labor group (Experimental): Pregnant women hospitalized for preterm labor
  Interventions: Other: lung and liver elastography measurement of fetus
- control group (Other): Pregnant women with a normal pregnancy
  Interventions: Other: lung and liver elastography measurement of fetus

INTERVENTIONS:
Other: lung and liver elastography measurement of fetus

SUMMARY:
The objective of the study was to evaluated the feasibility and reproducibility of the measurement of lung elasticity report / fetal liver according to gestational age in a group of patients with a normal course of pregnancy and in a group of Patients at risk of preterm delivery.

ELIGIBILITY:
Inclusion Criteria for control group :

* major pregnant women
* singleton pregnancy

Inclusion Criteria for control group :

* major pregnant women
* singleton pregnancy
* hospitalized for threatened premature birth between 24 and 34 WA
* Indication of a cure corticosteroid betamethasone

Exclusion Criteria:

* maternal conditions of pregnancy: diabetes gestational, pregnancy-induced hypertension, preeclampsia
* fetal lung diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Evolution over 48 hours of the fetal lung elasticity coefficient measure in kilopascals (kPa) (compared to the fetal liver) | For pretern larbor group: day of hospitalization for preterm labor, then 2 days later. For control group, both measurements at 2-day intervals
  The dates of elastography exams controls patients will be distributed a week of amenorrhea (WA) between 24 and 34 WA.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mottet N, Aubry S, Vidal C, Boiteux G, Metz JP, Riethmuller D, Pazart L, Ramanah R. Feasibility of 2-D ultrasound shear wave elastography of fetal lungs in case of threatened preterm labour: a study protocol. BMJ Open. 2017 Dec 26;7(12):e018130. doi: 10.1136/bmjopen-2017-018130. PMID 29282263